CLINICAL TRIAL: NCT05015192
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Single Ascending Dose of NH102 in Healthy Subjects
Brief Title: Single Ascending Dose Study of NH102 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Nhwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NH102-11
Record Dates: First submitted 2021-08-19; First posted 2021-08-20 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- NH102 3mg (Experimental): NH102 3mg, tablet, orally, once on Day 1 or NH102 placebo-matching tablet, orally, once on Day 1. NH102 or placebo will be administered after an overnight fast of approximately at least 10 hours.
  Interventions: Drug: NH102; Drug: Placebo
- NH102 9mg (Experimental): NH102 9mg, tablet, orally, once on Day 1 or NH102 placebo-matching tablet, orally, once on Day 1. NH102 or placebo will be administered after an overnight fast of approximately at least 10 hours.
  Interventions: Drug: NH102; Drug: Placebo
- NH102 20mg (Experimental): NH102 20mg, tablet, orally, once on Day 1 or NH102 placebo-matching tablet, orally, once on Day 1. NH102 or placebo will be administered after an overnight fast of approximately at least 10 hours.
  Interventions: Drug: NH102; Drug: Placebo
- NH102 40mg (Experimental): NH102 40mg, tablet, orally, once on Day 1 or NH102 placebo-matching tablet, orally, once on Day 1. NH102 or placebo will be administered after an overnight fast of approximately at least 10 hours.
  Interventions: Drug: NH102; Drug: Placebo
- NH102 60mg (Experimental): NH102 60mg, tablet, orally, once on Day 1 or NH102 placebo-matching tablet, orally, once on Day 1. NH102 or placebo will be administered after an overnight fast of approximately at least 10 hours.
  Interventions: Drug: NH102; Drug: Placebo
- NH102 80mg (Experimental): NH102 80mg, tablet, orally, once on Day 1 or NH102 placebo-matching tablet, orally, once on Day 1. NH102 or placebo will be administered after an overnight fast of approximately at least 10 hours.
  Interventions: Drug: NH102; Drug: Placebo

INTERVENTIONS:
Drug: NH102 — tablets, orally
  Other Names: H04
Drug: Placebo — tablets, orally

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics (PK) of NH102 when administered as single oral dose at escalating dose levels in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called NH102. NH102 is being tested to treat people who have depression. This study will look at the safety, tolerability and PK of NH102 in healthy participants.

The study may enroll up to 72 participants. Participants will be randomly assigned within each cohort to receive NH102 or placebo which will remain undisclosed to the participants and study doctor during the study (unless there is an urgent medical need). Each cohort will enroll 12 participants，which including 2 sentries (all were male, one receive NH102 and the other receive placebo) and 10 subjects(4 males and 4 females receive NH102 and 1 male and 1 female receive placebo). Participants enrolled in Cohort 1 to 6 will receive NH102 3mg, 9mg, 20mg, 40mg, 60mg and 80 mg or NH102 placebo-matching tablet. 2 sentries in all cohorts can be administered at the same time, and the remaining subjects of the same cohort can be administered only after observation for at least 24 hours and initial safety confirmation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 45 (both inclusive) years old when signing the informed consent.
2. Healthy volunteers has a body weight ≥50 kg (for male) or ≥ 45kg (for female) and body mass index ≥18.5 and ≤28 kg/m2 at screening.
3. Subjects voluntarily participate and sign the informed consent after understanding the purpose, content, procedures and possible risks of the trial.
4. The subjects will be able to communicate well with the investigators, be willing and able to comply with the lifestyle restrictions specified in the protocol, and cooperate to complete the study.

Exclusion Criteria:

1. The investigator determined that the subjects' present medical history and past medical history had any disease or dysfunction that would affect the clinical trial, including but not limited to diseases of the central nervous system, cardiovascular system, respiratory system, digestive system, urinary system, endocrine system, hematological system, etc.
2. There is any surgical condition or disease that may significantly affect the absorption, distribution, metabolism and excretion of drugs, or may harm to the subjects participating in the trial; such as history of gastrointestinal operations (gastrectomy, gastroenterostomy, enterectomy, etc.), urinary tract obstruction or dysuria, gastroenteritis, digestive tract ulcers, history of gastrointestinal bleeding, etc.
3. Subjects with past history of allergy to drugs or allergic disease.
4. Subjects with currently or past history of mental disorders and brain functional disorders.
5. According to the Columbia suicide severity scale (C-SSRS), subjects were at risk of suicide or were at risk of suicide based on the clinical judgment of the researchers, or with past history of self-injurious behavior.
6. Subjects have history of drug abuse or positive urine drug tests at screening within 1 year prior.
7. Subjects have history of alcohol abuse(i.e.,criteria are per week consumption more than 14 standard units(1 unit =360mL beer or 45mL 40% alcohol of Chinese liquor or 150mL wine)or positive alcohol breath tests at screening within 1 year prior.
8. Average amount of daily smoking>5 cigarettes at screening 3 months prior.
9. Those who have special requirements for food, cannot follow a uniform diet or have difficulty swallowing.
10. Female subjects who are pregnant and lactating ; and those who refuse to use effective non-drug contraceptive measures (such as abstinence, intrauterine device) or have planned to donate sperm or ovum throughout the study period and within 3 months after the end of the study.
11. Abnormal vital signs, lab and ECG indicators, as determined by the researcher, and clinically significant (e.g., male QTC > 450ms female > 470ms,corrected by Friericia ).
12. Subjects who resting heart rate <55 beats/min or >100 beats/min; systolic blood pressure <90mmHg or >140mmHg; diastolic blood pressure <60mmHg or >90mmHg.
13. Subjects who hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCV-Ab), or HIV antibody (HIV-Ab), or syphilis serum reaction (TRUST) is non-negative.
14. Subjects who participated in any clinical trial within 3 months before medication.
15. Subjects have history of blood donations of 400 mL within 3 months before enrollment; 200 mL within 1 month before enrollment; or have history of using blood products.
16. Subjects who had a history of surgery within 3 months prior to enrollment, or did not recover from surgery, or had an expected surgical plan during the study period.
17. Subjects who had taken any drugs, including prescription and over-the-counter drugs within 2 weeks prior to enrollment.
18. Subjects who directly related to this clinical trial.
19. Subjects have poor compliance or other problems that the researchers believe that it is not suitable for participating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Baseline up to Day 11
  To investigate the safety and tolerability of NH102 by assessment of AEs following administration in SAD

SECONDARY OUTCOMES:
PK parameters - Cmax | up to 72 hours
  Maximum Observed Plasma Concentration of NH102
PK parameters - Tmax | up to 72 hours
  Time to Reach the Maximum Plasma Concentration (Cmax) of NH102
PK parameters - AUC0-∞ | up to 72 hours
  area under the concentration versus time curve (AUC) from time zero to infinity
PK parameters - t½ | up to 72 hours
  apparent terminal elimination half-life
PK parameters - Vz/F | up to 72 hours
  apparent volume of distribution
PK parameters - CL/F | up to 72 hours
  the Apparent Clearance

CONTACTS AND LOCATIONS:
Overall Officials: Huafang Li, MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China